CLINICAL TRIAL: NCT04833140
Title: Estrogen Administration for the Treatment of NASH in Postmenopausal Women
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Chief, Neuroendocrine Unit, Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021P001506
Record Dates: First submitted 2021-04-03; First posted 2021-04-06 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Ortho Evra

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Estradiol (Active Comparator): Estradiol in the form of a transdermal patch 100 mcg daily (Vivelle-Dot generic).
  Women with an intact uterus will also receive progesterone (100 mg) in the form of a vaginal tablet (Endometrin, Ferring Pharmaceuticals, Inc.) inserted daily for endometrial protection
  Interventions: Drug: Estradiol patch
- Placebo (Placebo Comparator): Placebo patch (containing no estradiol) Women with an intact uterus will also receive vaginal placebo capsules (containing no progesterone)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estradiol patch — The patch will provide 100mcg of estradiol daily.
  Arms: Estradiol
Drug: Placebo — Placebo patch will contain no estradiol.
  Arms: Placebo

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a growing epidemic in the United States. Despite this, the treatment options remain limited. Preclinical and preliminary clinical data suggest that estrogen deficiency plays an important role in the pathology of steatosis, inflammation and fibrosis in non-alcoholic steatohepatitis (NASH), the progressive form of NAFLD. Post-menopausal women are a growing population with particularly high risk of NASH due to their lack of estrogen. This study will examine the effect of estradiol on hepatic fibrosis and fat in post-menopausal women with NASH.

ELIGIBILITY:
Inclusion criteria:

* Postmenopausal women 45-70 years old
* NASH by biopsy or NAFLD by imaging within 6 months of screen
* Hepatitis C antibody and hepatitis B surface antigen negative
* Negative mammogram within 1 year

Exclusion criteria:

* Heavy alcohol use
* Use of NASH pharmacotherapies within 12 months of study entry
* Known cirrhosis, stage 4 fibrosis on biopsy, or clinical evidence of cirrhosis or portal hypertension on imaging or exam
* Participation in NASH clinical trial within 6 months of study entry
* Chronic use of corticosteroids, methotrexate, amiodarone, or tamoxifen within 6 months of entry
* Known diagnosis of chronic liver disease other than NAFLD or found on biopsy
* Contraindication to liver biopsy including INR > 1.5, platelets < 50,000/mL, ascites, chronic anticoagulation (other than aspirin), biliary obstruction, peritonitis, inability to lie supine for 30 minutes
* Hgb < 10.0 g/dL or glomerular filtration rate < 60 mL/min
* Contraindications to estrogen therapy
* Any vaginal bleeding, including spotting, within the last year
* Active malignancy
* Severe chronic illness
* Use of estrogen or progesterone within a year of baseline visit
* Routine MRI exclusion criteria such as the presence of a pacemaker or cerebral aneurysm clip

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Liver fat | 12 months
  Reduction in amount of fat in the liver

CONTACTS AND LOCATIONS:
Overall Officials: Karen K. Miller, MD, Principal Investigator — Massachsuetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No